CLINICAL TRIAL: NCT04795752
Title: Prospective, Randomized, Masked, Controlled Trial To Evaluate The Safety And Effectiveness Of The TearCare® System In The Treatment Of The Signs And Symptoms Of Dry Eye Disease (SAHARA)
Brief Title: Safety And Effectiveness Of The TearCare® System In The Treatment Of The Signs And Symptoms Of Dry Eye Disease (SAHARA)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sight Sciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 07093
Record Dates: First submitted 2021-03-09; First posted 2021-03-12 (Actual); Results first posted 2025-11-24 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Dry Eye; Meibomian Gland Dysfunction
MeSH Terms: conditions — Dry Eye Syndromes; Meibomian Gland Dysfunction | interventions — Cyclosporins

STUDY DESIGN:
Intervention Model Description: Randomized parallel group through Month 6 (primary endpoint); TearCare arm continue follow-up through Month 24 to assess durability of treatment; Restasis arm stops Restasis at Month 6 and receives a single TearCare treatment then followed for an additional 6 months through Month 12. Extension portions for both arms are non-comparative.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (3):
- TearCare Group (Study Device) (Baseline to Month 24) (Experimental): TearCare System
  Interventions: Device: TearCare System
- Restasis Group (Control) (Baseline to Month 6) (Active Comparator): Restasis® (0.05% Cyclosporine ophthalmic emulsion).
  Interventions: Drug: Cyclosporine Ophthalmic 0.05% Ophthalmic Emulsion
- Restasis group crossed over to TearCare (Month 6 to Month 12) (Experimental): Subjects originally randomized to Restasis stop Restasis use at Month 6 and receive a single TearCare treatment at Month 6 and are then followed through Month 12.
  Interventions: Device: TearCare System

INTERVENTIONS:
Device: TearCare System — TearCare procedures in this study will include an in-office eyelid debridement, 15 minute bilateral thermal session with the TearCare System, immediately followed by manual expression of the meibomian glands using the Clearance Assistant Plus device. Subjects randomized to TearCare will receive one in-office TearCare procedure within 7 days of the Baseline visit and at 5 Months.
  Arms: Restasis group crossed over to TearCare (Month 6 to Month 12); TearCare Group (Study Device) (Baseline to Month 24)
Drug: Cyclosporine Ophthalmic 0.05% Ophthalmic Emulsion — Restasis group will be required to self-administer 1 drop twice a day from baseline through the Month 6 visit. At the Month 6 visit subjects will stop Restasis and receive a single TearCare treatment.
  Other Names: Restasis
  Arms: Restasis Group (Control) (Baseline to Month 6)

SUMMARY:
To demonstrate the safety and effectiveness of TearCare® procedures compared to Restasis® to treat the signs and symptoms of dry eye disease in adult patients.

DETAILED DESCRIPTION:
In this prospective, multicenter, randomized, active-controlled trial, TearCare is compared to cyclosporine 0.05% ophthalmic emulsion (Restasis) in eyes with dry eye disease (DED). Subjects randomized to TearCare receive TearCare treatment at baseline and Month 5, while subjects randomized to Restasis dose twice-daily with Restasis from baseline through Month 6. Primary inference is based on outcomes at the Month 6 visit including the co-primary endpoints tear break-up time (TBUT) and Ocular Surface Disease Index (OSDI).

ELIGIBILITY:
Inclusion Criteria:

* At least 22 years of age
* Reports dry eye symptoms within the past 3 to 6 months
* Reports having to use artificial tears or lubricants regularly over the past month to relieve dry eye symptoms.
* Schirmer tear test (with anesthesia) ≥1 to ≤10 mm in 5 minutes
* OSDI Score of 23-79
* TBUT of ≥1 to ≤7 seconds in both eyes
* Meibomian gland obstruction in both eyes based on a total Meibomian Gland Secretion Score ≤12 in each eye.
* At least 15 glands in each lower eyelid should be expressible, with a sterile cotton swab, at the slit lamp.
* Best corrected visual acuity of 20/100 or better in both eyes.
* Willing and able to comply with the study procedures and follow-up
* Willing and able to provide informed consent
* English-speaking

Exclusion Criteria:

* Use of any of the following medications:

  1. Cyclosporine (Restasis, Cequa etc.) or Xiidra within 60 days prior to enrollment;
  2. Antihistamines (oral or topical) within 10 days prior to enrollment;
  3. Systemic medication(s) (other than antihistamines) that is known to cause ocular dryness (e.g. diuretics, anti-hypertensives, anti-depressants, hormone therapy) and whose dose of this medication(s) has not been stable within 30 days prior to enrollment. There must be no anticipated adjustments to the dose of these medications for the duration of the trial;
  4. Accutane (at any time);
  5. Oral tetracyclines or azithromycin within 30 days prior to enrollment; or
  6. Topical ophthalmic antibiotics, anti-glaucoma medications, steroids, non-steroidal anti- inflammatory medications within 30 days prior to enrollment.
* Any of the following dry eye treatments:

  1. Office-based dry eye treatment (e.g. IPL, TearCare, thermal pulsation [Lipiflow], iLux etc.) within 12 months prior to enrollment either as part of routine care or clinical investigation;
  2. Meibomian gland expression within 6 months prior to enrollment;
  3. Blephex or debridement within 3 months prior to enrollment is an exclusion;
  4. Punctal occlusion or punctal plugs. Investigators can choose to remove the punctal plugs 15 days prior to enrollment;
  5. Use of TrueTear device within the past 2 weeks. (Subjects must refrain from using the TrueTear device for the duration of the study.); or
  6. Any history of meibomian gland probing
* History of eyelid, conjunctiva or corneal surgery (including refractive surgery) within the past year. In addition, subjects with any history of the following are excluded: chalazion surgery, surgery on the tarsal conjunctiva, radial keratotomy (RK), complicated blepharoplasty, lid reconstruction, or significant complications post-refractive surgery.
* Contact lens use within the past 2 weeks.
* History of Ocular Herpes Simplex or Ocular Herpes Zoster
* Any active, clinically significant ocular or peri-ocular infection or inflammation
* Recurrent clinically significant eye inflammation, other than dry eye, within 3 months prior to enrollment
* Clinically significant anterior blepharitis. In addition, collarettes or flakes of more than one quarter of the eyelid are excluded.
* Clinically significant eyelid abnormalities in either eye (e.g. entropion/ectropion, blepharospasm, aponeurotic ptosis, lagophthalmos, distichiasis, trichiasis).
* Clinically significant dermatologic or cutaneous disease of the eyelid or periocular area.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 345 (Actual)
Dates: Start 2021-04-28 (Actual); Primary Completion 2024-09-23 (Actual); Study Completion 2024-09-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jaime Dickerson, PhD, Study Director — Sight Sciences, Inc.
Locations (14):
- United States (14):
  - Doctor My Eyes, Scottsdale, Arizona
  - Scripps Health, La Jolla, California
  - Harvard Eye Associates, Laguna Hills, California
  - Eye Research Foundation, Newport Beach, California
  - Vision Institute, Colorado Springs, Colorado
  - Loh Ophthalmology Associates, Miami, Florida
  - Jackson Eye, Lake Villa, Illinois
  - Cincinnati Eye Institute, Edgewood, Kentucky
  - Kentucky Eye Institute, Lexington, Kentucky
  - Vita Eye Clinic, Shelby, North Carolina
  - Vantage Eye Care, Bala-Cynwyd, Pennsylvania
  - University of Pittsburg-Ophthalmology Dept, Pittsburgh, Pennsylvania
  - Vance Thompson Vision, Sioux Falls, South Dakota
  - Parkhurst NuVision, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hovanesian J, Ayres BD, Bloomenstein MR, Loh J, Chester T, Saenz B, Echegoyen J, Kannarr SR, Rodriguez TC, Dickerson JE Jr. Durability of the TearCare treatment effect in subjects with dry eye disease: Stage 3 of the Sahara randomized controlled trial. Optom Vis Sci. 2025 Aug 1;102(8):495-504. doi: 10.1097/OPX.0000000000002278. Epub 2025 Jul 25. PMID 40719437

RESULTS

PARTICIPANT FLOW:
Groups:
- TearCare Group (Study Device): TearCare System
  TearCare System: TearCare procedures in this study will include an in-office eyelid debridement, 15 minute bilateral thermal session with the TearCare System, immediately followed by manual expression of the meibomian glands using the Clearance Assistant Plus device. Subjects randomized to TearCare will receive one in-office TearCare procedure within 7 days of the Baseline visit and at 5 Months. Beginning at 9 Months, subjects will receive an additional TearCare procedure when TBUT drops lower than Baseline or within 2 seconds of baseline AND/OR if OSDI worsens by at least 1 category. These subjects will continue follow-up through 24 months.
- Restasis Group (Control): Restasis® (0.05% Cyclosporine ophthalmic emulsion
  Restasis: Restasis group will be required to self-administer 1 drop twice a day from baseline through the Month 6 visit. At Month 6, subjects will be crossed over to the TearCare group and will receive one (1) TearCare procedure. Following this single TearCare procedure, these subjects will be followed for an additional 6 months (12 months total).
Period: Primary Endpoint Phase
Arm/Group | TearCare Group (Study Device) | Restasis Group (Control)
Started | 172 | 173
Completed | 155 (Month 6 (primary endpoint) completion.) | 163 (Month 6 primary endpoint completion.)
Not Completed | 17 | 10
Not completed — Withdrawal by Subject | 7 | 7
Not completed — Lost to Follow-up | 3 | 2
Not completed — Physician Decision | 2 | 0
Not completed — Other | 4 | 1
Not completed — Protocol Violation | 1 | 0
Period: X-over-Restasis arm; Durability-TC arm
Arm/Group | TearCare Group (Study Device) | Restasis Group (Control)
Started | 155 | 163
Completed | 142 | 161
Not Completed | 13 | 2
Not completed — Lost to Follow-up | 7 | 0
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Physician Decision | 1 | 0
Not completed — Death | 1 | 0
Not completed — Other | 3 | 1

BASELINE CHARACTERISTICS:
Units Other Than Participants: eyes
Groups:
- TearCare Group (Study Device): TearCare System
  TearCare System: TearCare procedures in this study will include an in-office eyelid debridement, 15 minute bilateral thermal session with the TearCare System, immediately followed by manual expression of the meibomian glands using the Clearance Assistant Plus device. Subjects randomized to TearCare will receive one in-office TearCare procedure within 7 days of the Baseline visit and at 5 Months.
- Restasis Group (Control): Restasis® (0.05% Cyclosporine ophthalmic emulsion
  Restasis: Restasis group will be required to self-administer 1 drop twice a day from baseline through the Month 6 visit.
- Total: Total of all reporting groups
Arm/Group | TearCare Group (Study Device) | Restasis Group (Control) | Total
Number analyzed (Participants) | 172 | 173 | 345
Number analyzed (eyes) | 344 | 346 | 690
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 113 | 114 | 227
  >=65 years | 59 | 59 | 118
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.5 (14.8) | 56.8 (13.1) | 56.2 (14.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 120 | 128 | 248
  Male | 52 | 45 | 97
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Subject Demographics: Asian | 9 | 7 | 16
  Subject Demographics: Black/African American | 6 | 12 | 18
  Subject Demographics: White/Caucasian | 155 | 151 | 306
  Subject Demographics: Other/mixed | 2 | 3 | 5
Region of Enrollment [Number; unit: participants]
  United States | 172 | 173 | 345
Tear Break Up Time [Mean (Standard Deviation); unit: seconds] — Change in the measured time (in seconds) for the tear film to break up between baseline and Month 6. Measured for each eye of a subject.
  seconds | 4.39 (1.26) | 4.37 (1.18) | 4.38 (1.21)
OSDI [Mean (Standard Deviation); unit: units on a scale] — Change in Ocular Surface Disease Index (OSDI) between baseline and Month 6. OSDI is a scale ranging from 0 to 100, with a higher score indicating worse symptoms.
  units on a scale | 50.0 (14.9) | 50.0 (14.9) | 50.0 (14.9)

OUTCOME MEASURES:

1. Primary Outcome: Tear Break-Up Time
Description: Change in Tear Break-Up Time (TBUT) from baseline to month 6
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: seconds
Units Other Than Participants: eyes
Groups:
- TearCare Group (Study Device): TearCare System
  TearCare System: TearCare procedures in this study will include an in-office eyelid debridement, 15 minute bilateral thermal session with the TearCare System, immediately followed by manual expression of the meibomian glands using the Clearance Assistant Plus device. Subjects randomized to TearCare will receive one in-office TearCare procedure within 7 days of the Baseline visit and at 5 Months. Beginning at 9 Months, subjects will receive an additional TearCare procedure when TBUT drops lower than Baseline or within 2 seconds of baseline AND/OR if OSDI worsens by at least 1 category.
- Restasis Group (Control): Restasis® (0.05% Cyclosporine ophthalmic emulsion
  Restasis: Restasis group will be required to self-administer 1 drop twice a day from baseline through the Month 6 visit. At Month 6, subjects will be crossed over to the TearCare group and will receive one (1) TearCare procedure.
Arm/Group | TearCare Group (Study Device) | Restasis Group (Control)
Number analyzed (Participants) | 172 | 173
Number analyzed (eyes) | 344 | 346
seconds | 2.71 (3.35) | 1.22 (2.46)

2. Primary Outcome: OSDI Score
Description: Change in Ocular Surface Disease Index (OSDI) score from baseline to 6-months. The OSDI is a 12-item questionnaire that assesses symptoms of ocular irritation associated with dry eye and the impact of these on vision-related activities. The OSDI score ranges from 0 (best possible) to 100 (worst possible). The change in OSDI questionnaire from baseline to Month 6 is the difference between the scores at the two timepoints. A negative value would indicate improvement and a positive value, a worsening. The reported value is the mean of the change for all subjects.
Time Frame: 6 months
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | TearCare Group (Study Device) | Restasis Group (Control)
Number analyzed (Participants) | 172 | 173
score on a scale | -18.25 (17.98) | -15.53 (19.86)

ADVERSE EVENTS:
Time Frame: 24 months; TearCare subjects were followed for 24 months while Restasis subjects were followed for 12 months.
Description: AEs were monitored and collected for the Safety population - All subjects exposed to treatment.
Groups:
- TearCare Group (Study Device) (Baseline to 24 months): TearCare System
  TearCare System: TearCare procedures in this study will include an in-office eyelid debridement, 15 minute bilateral thermal session with the TearCare System, immediately followed by manual expression of the meibomian glands using the Clearance Assistant Plus device. Subjects randomized to TearCare will receive one in-office TearCare procedure within 7 days of the Baseline visit and at 5 Months; this arm followed through 24 months.
- Restasis Group (Control) (Baseline to Month 6): Restasis® (0.05% Cyclosporine ophthalmic emulsion
  Restasis: Restasis group will be required to self-administer 1 drop twice a day from baseline through the Month 6 visit.
- Restasis Subjects crossed over to TearCare (Month 6- Month 12: Subjects randomized to Restasis stopped Restasis at Month 6 and received a single TearCare treatment at Month 6. Subjects were followed through Month 12.
Arm/Group | TearCare Group (Study Device) (Baseline to 24 months) | Restasis Group (Control) (Baseline to Month 6) | Restasis Subjects crossed over to TearCare (Month 6- Month 12
All-Cause Mortality (participants affected / at risk) | 1/172 | 0/173 | 0/163
Serious Adverse Events (participants affected / at risk) | 2/172 | 0/173 | 0/163
Other Adverse Events (participants affected / at risk) | 23/172 | 15/173 | 8/163
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TearCare Group (Study Device) (Baseline to 24 months) (N=172) | Restasis Group (Control) (Baseline to Month 6) (N=173) | Restasis Subjects crossed over to TearCare (Month 6- Month 12 (N=163)
Cholelithiasis (General disorders) | 1 (1) | 0 (0) | 0
Pulmonary Edema (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0
Gall bladder tumor (Hepatobiliary disorders) | 1 (1) | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TearCare Group (Study Device) (Baseline to 24 months) (N=172) | Restasis Group (Control) (Baseline to Month 6) (N=173) | Restasis Subjects crossed over to TearCare (Month 6- Month 12 (N=163)
Eyelid irritation (Eye disorders) | 1 (1) | 0 (0) | 1 (1)
chalazion (Eye disorders) | 4 (4) | 1 (1) | 0 (0)
Foreign body sensation (Eye disorders) | 1 (1) | 2 (2) | 0 (0)
New Onset Vitreous Floaters and Photopsia (Eye disorders) | 0 (0) | 3 (3) | 1 (1)
Posterior vitreous detachment (Eye disorders) | 1 (1) | 1 (1) | 0 (0)
Preseptal Cellulitis (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Subconjunctival Hemorrhage (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Vitreomacular Traction (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Worsening of Dry Eye (Eye disorders) | 2 (2) | 0 (0) | 0 (0)
Worsening of Preexisting condition (Eye disorders) | 0 (0) | 0 (0) | 1 (1) — glaucoma
Infection eyelid or ocular surface (Eye disorders) | 1 (1) | 0 (0) | 0 (0) — viral conjunctivitis
Loss of BCVA of ≥ 10 letters (Eye disorders) | 6 (7) | 2 (4) | 4 (4)
Swelling of the eyelid(s) (Eye disorders) | 2 (2) | 0 (0) | 0 (0)
Allergic Conjunctivitis (Eye disorders) | 1 (1) | 1 (1) | 0 (0)
Blepharitis (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Blurred Vision (Eye disorders) | 1 (1) | 1 (1) | 0 (0)
Conjunctival hyperemia (Eye disorders) | 1 (1) | 1 (1) | 0 (0)
Corneal Erosion (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Discomfort post instillation of drops (Eye disorders) | 0 (0) | 2 (2) | 0 (0)
conjunctival cyst (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Filamentary keratitis (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
blepharochalasis (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
macular degeneration (Eye disorders) | 2 (2) | 0 (0) | 0 (0)
canaliculitis (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
corneal infiltrate (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
epiretinal membrane (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
macular cystic changes (Eye disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After Sponsor's publication of trial results, the Institution and Principal Investigator may publish the results of the Study generated by the Institution, subject to the obligations of the CTA, and prior approval of Sponsor in writing. The Institution shall furnish Sponsor with a written copy of any proposed publication or disclosure at least 60 days prior to submission for publication or disclosure. Sponsor may request changes or other measures to ensure the information is fairly stated.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-08-26): https://cdn.clinicaltrials.gov/large-docs/52/NCT04795752/Prot_SAP_001.pdf